CLINICAL TRIAL: NCT05282576
Title: Effect of Neurophysiological Facilitation Techniques on Functional Levels and Respiratory in Intensive Care Patients
Brief Title: Effect of Neurophysiological Facilitation Techniques in Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Medical Park Hospital Istanbul (Other)
Responsible Party: Principal Investigator, Mehmet Burak Uyaroğlu, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Saglik Bilimleri Uni
Record Dates: First submitted 2022-02-26; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Intensive Care (ICU) Myopathy; Intensive Care Unit Acquired Weakness
Keywords: Intensive Care Unit; Critical Ill; Physiotherapy; Neurophysiologic Facilitation Techniques; Intensive Care Unit Acquired Weakness
MeSH Terms: conditions — Muscular Diseases | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Active Comparator): We applied neurophysiological facilitation techniques in addition to conventional rehabilitation.
  Interventions: Other: NPF Group
- Control Group (Other): Critical ill patients was applied their conventional physiotherapy
  Interventions: Other: Control Group

INTERVENTIONS:
Other: NPF Group — Participants allocated to the experimental group completed until discharged, neurophysiological facilitation(NPF) techniques in addition to conventional physiotherapy.
  Other Names: Neurophysiological facilitation techniques in addition to conventional physiotherapy.
  Arms: Experimental Group
Other: Control Group — Critical ill patients was applied their conventional physiotherapy which includes chest physiotherapy and mobilization until discharged
  Other Names: Conventional physiotherapy
  Arms: Control Group

SUMMARY:
The aim of this study was to investigate the effect of neurophysiological facilitation techniques on respiratory and functional levels in intensive care patients. Participants were divided into two groups as experimental (n=20) and control (n=20). Conventional physiotherapy, which includes chest physiotherapy, mobilization exercises and range of motion exercises were applied in control group. Neurophysiological facilitation techniques in addition to the conventional physiotherapy program ere applied in experimental group. The functional status, lower and upper extremity muscle strength, grip strength measurements of the patients and the rates of weaning from mechanical ventilation were evaluated before and after treatment. Vital signs, dyspnea and fatigue perception were assessed each day of treatment. Evaluations were analyzed statistically using Statistical Package for the Social Sciences-22 program.

DETAILED DESCRIPTION:
The intensive care unit is a multidisciplinary unit in which patients with acute, life-threatening organ dysfunction or under risk are monitored and treated comprehensively. Advanced technology is used for follow-up and treatment in intensive care. These supports decrease the mortality rate. However, the increase length of stay in the ICU leads to higher hospital costs in addition to serious secondary pathologies. Prolonged immobilisation in the intensive care unit(ICU); causes the loss of muscle mass and strength of the patients. When the course of illness, the medical devices used, various medications, malnutrition and other reasons such as sepsis are accompanied by this immobilization, the disorder called Intensive Care Acquired Muscle Weakness (ICU-AW) occurs. This neuromuscular disorder, also causes functional impairments after ICU discharge.

Early physiotherapy intervention in ICU, has a positive effect on the symptoms frequently occur in patients. In addition to improve the functional status of the patient such as exercise capacity, muscle strength and mobilization, its increase weaning from mechanical ventilation, and decrease the length of stay in the ICU and hospital. It also provides airway clearance, reduction the work of breathing and improvement of respiratory function.

Neurophysiological facilitation of respiration is the use of proprioceptive and tactile stimulation that produce reflexive movement responses. These responses provide to increase the depth of breathing, decrease respiratory rate in patients with decreased level of consciousness. It also increase inspiratory expansion of the ribs, epigastric excursion and abdominal muscles tone. In the study conducted Kumar et al. has indicated that neurophysiological facilitation (NPF) techniques improves levels of dyspnea and oxygen saturation (spO2) in Coronavirus patients. It is very important to increase the level of oxygen saturation to rate the mortality. In NPF techniques, respectively the proprioceptors and tactile receptors in the abdominal, intercostals and spinal muscles are affected, phrenic motor neurons are stimulated, thoracic and abdominal excursions are increased and thus provide improves vital parameters.

ELIGIBILITY:
Inclusion Criteria:

* Clinically Unstable
* Participants Over the Age of 18
* Individuals who volunteered to participate in the study or were allowed by their first-degree relatives if they were unconscious.
* Patients who are suitable for physiotherapy by the intensive care specialist.

Exclusion Criteria:

* Having coagulation disorder (INR > 1,5 platelet<50.000 mm3)
* Having neuromuscular diseases
* Having psychiatric disease or overly agitated (Richmond Agitation Sedation Scale score ≥ +2)
* Having acute stroke
* Having Raised Intracranial Pressure Syndrome symptoms
* Having cardiac and respiratory instability (Respiratory frequency > 30 breaths/min,Partial pressure of oxygen(PaO₂)< 65 mmHg , fraction of inspired oxygen(FiO₂)>%55, Diastolic blood pressure < 50 mmHg or > 200 mmHg , Systolic blood pressure < 80 mmHg or > 200 mmHg)
* Having hemodynamic instability (intropin dose > 5 mcg/kg/min)
* Fever
* Malignity
* Shock
* Patients admitted to ICU after cardiac, trauma and surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
The Chelsea Critical Care Physical Assessment Tool | through study completion, an average of 5 days
  The Chelsea Critical Care Physical Assessment Tool (CPAx) is a test used on male and female patients in the intensive care unit (ICU) to assess physical and respiratory function impairments and morbidity. The CPAx assessment also identifies patients at risk for developing ICU-acquired complications, such as weakness and mobility decline. The CPAx assesses 10 domains including respiratory function, cough, bed mobility, supine to sitting on edge of bed, dynamic sitting, standing balance, sit to stand, transferring bed to chair, stepping, and grip strength.
Physical Function in Intensive Care Test | through study completion, an average of 5 days
  Physical Function in Intensive Care Test(PFIT) is specifically for the patient population in the intensive care unit (ICU) who are critically ill. This test can be used to guide exercise prescription within the ICU as well as measure functional recovery. The PFIT-s is a battery outcome measure involving four components: sit to stand assistance, marching on the spot cadence, shoulder flexor and knee extensor strength. The PFIT include 4 items.
Premorbid Level of Activity Scales | through study completion, an average of 5 days
  Premorbid dyspnea was scored according to the American Thoracic Society (ATS) scale. The activities of daily living were recorded as 0 = working; 1 = independent (fully ambulatory and living without any assistance); 2 = restricted (able to live on their own and leave their homes to perform basic tasks, but severally limited in exercise ability); 3 = housebound (cannot leave their homes unassisted or leave their homes rarely, able to perform self-care but unable to do heavy chores such as house cleaning, cannot live alone, and may be institutionalized; and 4 = bedridden or wheelchair-bound

SECONDARY OUTCOMES:
Change in Heart Rate | During ICU stay
  Heart rate can be quantified easily at the bedside, while preload estimation has traditionally relied on invasive pressure measurements, both central venous and pulmonary artery wedge
Change in Blood Pressure | During ICU stay
  BP can be measured non-invasively using a sphygmomanometer (BP cuff).
Change in Oxygen saturation | During ICU stay
  Pulse oximetry is the technique used to measure arterial oxygen saturation in the peripheral blood vessels
Change in Respiratory Frequency | During ICU stay
  The respiratory frequency is usually measured when a person is at rest and simply involves counting the number of breaths for one minute by counting how many times the chest rises.
Change in Perception of Fatigue | During ICU stay
  the Perception of Fatigue is was assess to used The Borg Rating of Perceived Exertion(RPE). The Borg RPE scale is a numerical scale that ranges from 6 to 20, where 6 means "no fatigue at all" and 20 means "maximal fatigue.
Change in Perception of Dyspnea | During ICU stay
  the Perception of Dyspnea is was assess to used The Borg Rating of Perceived Exertion(RPE). The Borg RPE scale is a numerical scale that ranges from 6 to 20, where 6 means "no dyspnea at all" and 20 means "maximal dyspnea'.
The Functional Independence Measure | through study completion, an average of 5 days
  The The Functional Independence Measure (FIM) is an 18-item instrument measuring a person's level of disability in terms of burden of care. The FIM should be rated by the consensus opinion of a multidisciplinary team, but the evaluation is often performed by a single professional. Each item is rated from 1 (requiring total assistance) to 7 (completely independent). Three independent FIM scores can be generated by summing item scores: a total score (FIM total: 18 items), a motor score (FIM motor: eating, grooming, bathing, dressing - upper body, dressing - lower body, toileting, bladder management, bowel management, and transfers bed/chair/wheelchair, toilet, tub/shower, walk, stairs), and a cognitive score (FIM cognitive: auditory comprehension, verbal expression, social interaction, problem solving, and memory).
Change in Muscle Strength | through study completion, an average of 5 days
  Change in muscle strength was measured with a Digital Manual Muscle Tester.
Change in Hand Grip Strength | through study completion, an average of 5 days
  Change in Hand Grip Strength was measured with a Hydraulic Hand Dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Burak Uyaroğlu, PT,PhD, Study Director — Saglik Bilimleri Universitesi; Yasemin Çırak, Ass.Prof, Principal Investigator — Istinye University
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No